CLINICAL TRIAL: NCT03753477
Title: An Open-label, Randomized, 2X2 Crossover Study to Compare the Pharmacokinetics and Safety Between DWJ1351 and Co-administration of Amlodipine/Olmesartan and Rosuvastatin in Healthy Male Subjects
Brief Title: Clinical Trial to Investigate the Efficacy and Safety of DWJ1351
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1351004
Record Dates: First submitted 2018-02-14; First posted 2018-11-27 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Amlodipine; olmesartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Drug (Experimental): DWJ1351(FDC Amlodipine/Olmesartan/Rosuvastatin)
  Interventions: Drug: DWJ1351(FDC Amlodipine/Olmesartan/Rosuvastatin)
- Reference Drug (Active Comparator): Sevikar and Crestor
  Interventions: Drug: Sevikar and Crestor

INTERVENTIONS:
Drug: DWJ1351(FDC Amlodipine/Olmesartan/Rosuvastatin) — DWJ1351(FDC Amlodipine/Olmesartan/Rosuvastatin) X 1 tablet followed by Sevikar(Amlodipine/Olmesartan) X 1 tablet and Crestor(Rosuvastatin) X 1 tablet (after washout period)
  Other Names: DWJ1351
  Arms: Test Drug
Drug: Sevikar and Crestor — Sevikar(Amlodipine/Olmesartan) X 1 tablet and Crestor(Rosuvastatin) X 1 tablet followed by FDC Amlodipine/Olmesartan/Rosuvastatin X 1 tablet (after washout period)
  Other Names: Amlodipine/Olmesartan and Rosuvastatin
  Arms: Reference Drug

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetic characteristics of combination of amlodipine, olmesartan and rosuvastatin and DWJ1351 in healthy male volunteers

DETAILED DESCRIPTION:
The purpose of this study is to compare the safety and pharmacokinetic characteristics of combination of amlodipine, olmesartan and rosuvastatin and DWJ1351 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject who provided written informed consent to participate in this study
* Healthy adult male subjects aged 19 to 50 years
* Subjects whose body weight ≥ 55 kg and Body Mass Index(BMI) ≥ 18.0 kg/m2 and ≤ 27.0 kg/m2
* Subject who was judged to be healthy and suitable for the participation by the investigator based on screening test results

Exclusion Criteria:

* Subject who had a severe allergy or allergic reactions to the amlodipine, olmesartan, rosuvastatin or related drugs
* Subjects who had a serious clinical illness that can impact fate of drugs absorption
* Subject who shows vital signs with the number of systolic blood pressure of >140 mmHg or <100 mmHg, and the number of diastolic blood pressure of >90mmHg or <65mmHg
* Subject who have experienced drug abuse
* Subject who donates his blood (whole blood donation within last 2 months or plasma donation within last 1 month)
* Subject who has taken other clinical or licensed medication from another clinical trial within an 3-month period prior to the first administration of the study medication

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
AUC | [ Time Frame: 0 - 72 hours ]
  AUC
Cmax | [ Time Frame: 0 - 72 hours ]
  Cmax

SECONDARY OUTCOMES:
AUCinf | [ Time Frame: 0 - 72 hours ]
  AUCinf
Tmax | [ Time Frame: 0 - 72 hours ]
  Tmax
t1/2β | [ Time Frame: 0 - 72 hours ]
  t1/2β
CL/F | [ Time Frame: 0 - 72 hours ]
  CL/F
Vdss/F | [ Time Frame: 0 - 72 hours ]
  Vdss/F

CONTACTS AND LOCATIONS:
Overall Officials: JG Shin, Ph.D, Principal Investigator — Busan Paik Hospital
Locations (1):
- Busan Paik Hospital, Busan, South Korea